CLINICAL TRIAL: NCT04225260
Title: A Multicenter, Open-Label Study to Evaluate the Safety of QM1114-DP for the Long-term Treatment of Moderate to Severe Glabellar Lines and Lateral Canthal Lines
Brief Title: Long-term Treatment of Moderate to Severe Glabellar Lines and Lateral Canthal Lines
Acronym: READY-4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 43QM1903
Record Dates: First submitted 2020-01-07; First posted 2020-01-13 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2020-07

CONDITIONS: Glabellar Lines; Lateral Canthal Lines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- QM1114-DP in the LCL and the GL areas (Experimental): The investigational product (QM1114-DP) is a BoNT Type A.
  At each treatment a total dose of QM1114-DP will be administered in the glabella and lateral canthal lines.
  Interventions: Biological: botulinum toxin neuromodulator

INTERVENTIONS:
Biological: botulinum toxin neuromodulator — A dose of QM1114-DP will be injected in the GL area and in the LCL area.
  Other Names: QM1114-DP

SUMMARY:
This is a phase 3, multicenter, open-label study to evaluate the safety of QM1114-DP for the long term treatment of moderate to severe Glabellar (Frown) Lines (GL) and Lateral Canthal Lines (Crow's Feet and LCL).

ELIGIBILITY:
Inclusion Criteria:

- Male or female at least 18 years of age.

Exclusion Criteria:

* Previous use of any Botulinum toxin in facial areas within 9 months prior to study treatment.
* Anticipated need for treatment with botulinum toxin of any serotype for any reason during the study (other than the investigational product).
* Female who is pregnant, breast feeding, or intends to conceive a child during the study.
* Known allergy or hypersensitivity to any component of the investigational product (QM1114-DP) or any botulinum toxin serotype.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2021-04-12 (Actual); Study Completion 2021-05-21 (Actual)

CONTACTS AND LOCATIONS:
Locations (30):
- United States (29):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Investigate MD, LLC., Scottsdale, Arizona
  - Center for Dermatology Clinical Research, Inc., Fremont, California
  - Rejuva Medical Aesthetics, LLC, Los Angeles, California
  - Westside Aesthetics, Los Angeles, California
  - Marcus Facial Plastic Surgery, Redondo Beach, California
  - The Maas Clinic Research Center, San Francisco, California
  - ArteMedica, Santa Rosa, California
  - AboutSkin Research, LLC, Greenwood Village, Colorado
  - Modern Dermatology PC, Westport, Connecticut
  - Center for Clinical and Cosmetic Research, Aventura, Florida
  - Steven Fagien, MD, PA, Boca Raton, Florida
  - Susan H. Weinkle, M.D, Bradenton, Florida
  - Miami Skin and Vein LLC, Coral Gables, Florida
  - Mayoral Dermatology, Coral Gables, Florida
  - Skin Research Institute, LLC, Coral Gables, Florida
  - Research Institute of SouthEast, LLC, West Palm Beach, Florida
  - Hamilton Research LLC, Alpharetta, Georgia
  - Chicago Cosmetic Surgery and Dermatology, Inc, Chicago, Illinois
  - Pure Dermatology, LLC, Metairie, Louisiana
  - SkinCare Physicians, Chestnut Hill, Massachusetts
  - Skin Laser and Surgery Specialist of NY/NJ, Hackensack, New Jersey
  - Elite Aesthetic Research, Cincinnati, Ohio
  - Aventiv Research, Inc., Dublin, Ohio
  - Dallas Plastic Surgery Institute, Dallas, Texas
  - Center for Advanced Clinical Research, Dallas, Texas
  - Austin Institute for Clinical Research, Inc., Pflugerville, Texas
  - SkinDC, PLLC, Arlington, Virginia
  - EthiQ2 Research, LLC, Mequon, Wisconsin
- Jose Raul Montes Eyes & Facial Rejuvenation LLC, San Juan, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Groups:
- QM1114-DP in the LCL and the GL Areas: The investigational product (QM1114-DP) is a BoNT Type A.
  At each treatment a total dose of QM1114-DP will be administered in the glabella and lateral canthal lines.
  botulinum toxin neuromodulator: A dose of QM1114-DP will be injected in the GL area and in the LCL area.
Period: Overall Study
Arm/Group | QM1114-DP in the LCL and the GL Areas
Started | 902
Completed | 790
Not Completed | 112

BASELINE CHARACTERISTICS:
Arm/Group | QM1114-DP in the LCL and the GL Areas
Number analyzed (Participants) | 902
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.2 (11.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 775
  Male | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 12
  Native Hawaiian or Other Pacific Islander | 5
  Black or African American | 26
  White | 820
  More than one race | 16
  Unknown or Not Reported | 22
Region of Enrollment [Number; unit: participants]
  United States | 902

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieve Grade/Level 0 or 1 on the GL Investigator Scales at Maximum Frown
Description: 4-point scale
Time Frame: Week 4
Population: FAS
Measure: Count of Participants; unit: Participants
Groups:
- QM1114-DP in the GL: The investigational product (QM1114-DP) is a BoNT Type A.
  At each treatment a total dose of QM1114-DP will be administered in the glabella and lateral canthal lines.
  botulinum toxin neuromodulator: A dose of QM1114-DP will be injected in the GL area and in the LCL area.
Arm/Group | QM1114-DP in the GL
Number analyzed (Participants) | 847
Participants | 769

2. Primary Outcome: Percentage of Subjects Who Achieve Grade/Level 0 or 1 on the LCL Investigator Scales at Maximum Smile
Description: 4-point scale
Time Frame: Week 4
Measure: Count of Participants; unit: Participants
Groups:
- QM1114-DP in the LCL: The investigational product (QM1114-DP) is a BoNT Type A.
  At each treatment a total dose of QM1114-DP will be administered in the glabella and lateral canthal lines.
  botulinum toxin neuromodulator: A dose of QM1114-DP will be injected in the GL area and in the LCL area.
Arm/Group | QM1114-DP in the LCL
Number analyzed (Participants) | 847
Participants | 719

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | QM1114-DP in the LCL and the GL Areas
All-Cause Mortality (participants affected / at risk) | 1/902
Serious Adverse Events (participants affected / at risk) | 23/902
Other Adverse Events (participants affected / at risk) | 243/902
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QM1114-DP in the LCL and the GL Areas (N=902)
Appendicitis (Infections and infestations) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1)
Post procedural infection (Infections and infestations) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Urosepsis (Infections and infestations) | 1 (1)
Abdominal Pain Upper (Gastrointestinal disorders) | 1 (1)
Gastric ulcer (Gastrointestinal disorders) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1)
Adnocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
Cubital tunnel syndrome (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Post procedural hemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Goitre (Endocrine disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Trigger finger (Musculoskeletal and connective tissue disorders) | 1 (1)
Suicide (Psychiatric disorders) | 1 (1)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertensive urgency (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | QM1114-DP in the LCL and the GL Areas (N=902)
Injection site Pain (General disorders) | 65 (145)
Injection site bruising (General disorders) | 59 (71)
COVID-19 (Infections and infestations) | 48 (49)
Upper respiratory tract infection (Infections and infestations) | 15 (15)
Urinary Tract Infection (Infections and infestations) | 15 (16)
Sinusitis (Infections and infestations) | 9 (10)
Headache (Nervous system disorders) | 54 (56)
Alanine aminotransferase increased (Investigations) | 16 (16)
Aspartate aminotransferase increased (Investigations) | 15 (15)
Gamma-glutamyltransferase increased (Investigations) | 10 (10)
Hypertension (Vascular disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT04225260/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-05): https://cdn.clinicaltrials.gov/large-docs/60/NCT04225260/SAP_001.pdf